CLINICAL TRIAL: NCT01052727
Title: DOLCE Study: Day-care Versus Overnight-stay Laparoscopic Cholecystectomy Randomized, Controlled Trial
Brief Title: Day-care Versus Overnight-stay Laparoscopic Cholecystectomy Randomized Controlled Trial.
Acronym: DOLCE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal investigator: Dott. Luca Ansaloni, St. Orsola Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-DOLCE-01-2010-BO
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cholelithiasis
Keywords: Laparoscopic Cholecystectomy; quality of life
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- overnight stay group (Other): Group of patients who rests at least one night in Hospital
  Interventions: Procedure: Laparoscopic Cholecystectomy
- day-care Group (Other): Group of patients who is discharged tha same day of operation
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy

SUMMARY:
DOLCE Study: Day-care versus Overnight-stay Laparoscopic Cholecystectomy randomized, controlled trial.

The aim of this study was to evaluate the feasibility, safety and patient acceptance of outpatient LC in Italy. In particular this randomized clinical trial will use the SF-36 as powerful instrument to compare quality of life and global health status after LC performed as a day-care procedure or with an overnight stay.

Particular attention is taken to answer to the following methodological issues:

* concealed randomization,
* ITT analysis,
* number of eligible, excluded and refusing patients clearly stated.

DETAILED DESCRIPTION:
The DOLCE study project is a prospective, randomised, open label, comparison of LC performed either as a day-care procedure or with overnight stay with symptomatic gallstones.

The aim of this study was to evaluate the feasibility, safety and patient acceptance of outpatient LC in Italy. In particular this randomized clinical trial will use the SF-36 as powerful instrument to compare quality of life and global health status after LC performed as a day-care procedure or with an overnight stay.

The outcome measured are the following:

1. quality of life and health status
2. admissions and readmissions;
3. postoperative pain (SVS, number of analgesic doses);
4. wound infections (rate);
5. intraoperative and postoperative complications
6. duration of operation (minutes), defined as operating time, anesthesia time, or operating room time;
7. return to normal activity (days), subdivided in: time until return to full activity, work, or sport; The instrument used to assess quality of life and heath status will be SF-36. The study will be performed in a Day-Surgery Unit where an over-night stay is possible in case of complications.

INCLUSION AND EXCLUSION CRITERIA

Inclusion criteria are:

• Adult (from 18 to 70 years old) patients presenting for gallstone disease surgery (symptomatic cholelithiasis, according to the Rome criteria ) confirmed by ultrasound living less than 50 km from the hospital (the day-care protocol specifies that an adult must be available to accompany the patient home and stay there overnight) were considered for entry into the trial.

Exclusion criteria

* Refusing of informed consent
* Any condition preventing a correct evaluation of pain (non-cooperative patient, blind patient)
* Patients with contraindication to be operated with LC
* Patients with an American Society of Anesthesiologists (ASA) score of III or more.
* BMI >35 kg/m2
* Asthma
* extensive previous abdominal surgery
* patients with a clinical suspicion of common bile duct stones or a history of acute cholecystitis or pancreatitis, calcified gallbladder.

ELIGIBILITY:
Inclusion Criteria:

* Adult (from 18 to 70 years old) patients presenting for gallstone disease surgery (symptomatic cholelithiasis, according to the Rome criteria ) confirmed by ultrasound living less than 50 km from the hospital (the day-care protocol specifies that an adult must be available to accompany the patient home and stay there overnight) were considered for entry into the trial.

Exclusion Criteria:

* Refusing of informed consent
* Any condition preventing a correct evaluation of pain (non-cooperative patient, blind patient)
* Patients with contraindication to be operated with LC
* Patients with an American Society of Anesthesiologists (ASA) score of III or more.
* BMI >35 kg/m2
* Asthma
* extensive previous abdominal surgery
* patients with a clinical suspicion of common bile duct stones or a history of acute cholecystitis or pancreatitis, calcified gallbladder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
Evidence of better quality of life revealed by SF-36 test | before surgery, 7 days after surgery, 30 days after surgery

SECONDARY OUTCOMES:
Readmissions, Postoperative pain, Wound infections, Intraoperative and postoperative complications, Duration of operation(minutes), Return to normal activity (days) defined as time until return to full activity, work, school or sport. | prior to surgery, 7 days after surgery and 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St Orsola-Malpighi Hospital - University of Bologna, Bologna, Italy

REFERENCES:
- [Background] Ahmad NZ, Byrnes G, Naqvi SA. A meta-analysis of ambulatory versus inpatient laparoscopic cholecystectomy. Surg Endosc. 2008 Sep;22(9):1928-34. doi: 10.1007/s00464-008-9867-2. Epub 2008 Apr 9. PMID 18398648
- [Background] Gurusamy K, Junnarkar S, Farouk M, Davidson BR. Meta-analysis of randomized controlled trials on the safety and effectiveness of day-case laparoscopic cholecystectomy. Br J Surg. 2008 Feb;95(2):161-8. doi: 10.1002/bjs.6105. PMID 18196561